CLINICAL TRIAL: NCT04585087
Title: The Effect of Length of Adaptation on Threonine Requirement in Healthy Adult Men
Brief Title: Length of Adaptation and Threonine Requirement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Glenda Courtney-Martin, Health Systems Research Scientist, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1000071242
Record Dates: First submitted 2020-10-06; First posted 2020-10-14 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2021-10

CONDITIONS: Healthy
Keywords: Healthy; Adult; Men; Threonine; Dietary Requirement
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1 | interventions — Eating

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy adult men (Experimental): Participants will initially be seen for a pre-study assessment (2 hours). They will then be studied for up to 6 times (6 different levels of threonine intake). Each set of experiments will be 9-days in length. During the first 2 days, a pre-adaptation (milkshake) diet will be consumed. For the remaining 7 days, a protein liquid drink and protein-free cookies will be consumed. All of the diets will be provided by the investigators.
  During each 9-day experiment, participants are expected to come to the Clinical Research Centre at the Hospital for Sick Children for breath and urine collection (5 hours total for each visit)
  Interventions: Other: Dietary Intakes

INTERVENTIONS:
Other: Dietary Intakes — 6 levels of threonine intake will be provided by the protein liquid drink

SUMMARY:
This study aims to determine if the body's needs for threonine (an amino acid which is an essential building block for protein) is different when assessed after 1, 3 or 6 days of adaptation to the level of threonine intake being studied.

DETAILED DESCRIPTION:
Our method, the Indicator Amino Acid Oxidation (IAAO) method has been used before to look at amino acid requirements. Over the years, we have changed our method to make our studies on amino acid requirements safer to use in specific vulnerable populations like babies or older adults. For example, we have shown that we only need to collect breath and urine samples instead of collecting blood.

Another feature of our method is that we require subjects to consume personalized diets for 3 days at a time, repeated for up to 7 times. These personalized diets are important as they allow us to study the amount of amino acids needed by the body. The body's metabolism changes with different intakes of amino acids. We measure this change in metabolism by collecting breath and urine samples on the 3rd day of each diet period. However, we do not know if this specific length of time for the personalized diets (i.e. 3 days) is sufficient or whether more time is needed for the body to adjust to the amount of amino acids provided. There is a possibility that 3 days is not enough time and our results (i.e. our estimates of amino acid needs) may be different if we allow more time.

The purpose of this study is to find out if the threonine requirement determined using IAAO in adult men changes if the length of time on the personalized diets increases from 3 days to 5 and 9 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult men, 19 to 35 years of age
* Willingness to participate in the study and completed the screening procedures (height, weight, fasting blood sample and medical history questionnaire).
* No recent history of weight loss
* BMI between 18.5 - 27 kg/m 2
* Absence of chronic disease or acute illness that could affect protein and AA metabolism (diabetes, cancer, liver or kidney disease, HIV, acute cold or flu, hypo or hyperthyroidism, rheumatoid arthritis treated with anti-inflammatory medications).
* Non-smoking
* Willingness to consume the diet provided for 9 days

Exclusion Criteria:

1. Presence of disease known to affect protein and AA metabolism (diabetes, cancer, liver or kidney disease, HIV, acute cold or flu, hypo or hyperthyroidism, rheumatoid arthritis treated with anti-inflammatory medications).
2. On medications known to affect protein and amino acid metabolism (steroids).
3. Recent significant weight loss. ≥ 5% of body with in the last 3 months.
4. Individuals on weight reducing diets.
5. Inability to tolerate the diet
6. Unwilling to have blood drawn from a venous access, or using a ventilated hood indirect calorimeter for the purposes of the study.
7. Significant coffee consumption of more than 2 cups/day
8. Significant alcohol consumption of more than one drink/day
9. Failure to disclose any of the information needed to assess eligibility.

Ages: 19 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Determination of threonine requirement in young adult men after 8 hours, 3, and 7 days of adaptation to experimental diets. | 3 years
  The threonine requirement will be determined using IAAO and breakpoint analysis after 3 different lengths of adaptation to the experimental diet

CONTACTS AND LOCATIONS:
Overall Officials: Glenda Courtney-Martin, PhD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Szwiega S, Pencharz PB, Ball RO, Xu L, Kong D, Elango R, Courtney-Martin G. Length of Adaptation Has No Effect on the Threonine Requirement Determined in Healthy Young Adult Males Using the Indicator Amino Acid Oxidation Method. J Nutr. 2023 Jul;153(7):2016-2026. doi: 10.1016/j.tjnut.2023.03.033. Epub 2023 Mar 31. PMID 37004875